CLINICAL TRIAL: NCT00004260
Title: Phase I Study of Interleukin-12 in Combination With Rituximab in Patients With Non-Hodgkin's Lymphoma
Brief Title: Interleukin-12 Plus Rituximab in Treating Patients With Non-Hodgkin's Lymphoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Stephen Maxted Ansell, M.D., Mayo Clinic Cancer Center
Purpose: Treatment
Other Study IDs: CDR0000067514; U01CA069912 (NIH); 980112 (Other: Mayo Clinic Cancer Center)
Record Dates: First submitted 2000-01-28; First posted 2004-06-18 (Estimated); Last update posted 2011-08-03 (Estimated); Status verified 2011-08

CONDITIONS: Lymphoma
Keywords: stage I grade 1 follicular lymphoma; stage I grade 2 follicular lymphoma; stage I grade 3 follicular lymphoma; stage I adult diffuse small cleaved cell lymphoma; stage I adult diffuse mixed cell lymphoma; stage I adult diffuse large cell lymphoma; stage I adult immunoblastic large cell lymphoma; stage I adult lymphoblastic lymphoma; stage I adult Burkitt lymphoma; stage III grade 1 follicular lymphoma; stage III grade 2 follicular lymphoma; stage III grade 3 follicular lymphoma; stage III adult diffuse small cleaved cell lymphoma; stage III adult diffuse mixed cell lymphoma; stage III adult diffuse large cell lymphoma; stage III adult immunoblastic large cell lymphoma; stage III adult lymphoblastic lymphoma; stage III adult Burkitt lymphoma; stage IV grade 1 follicular lymphoma; stage IV grade 2 follicular lymphoma; stage IV grade 3 follicular lymphoma; stage IV adult diffuse small cleaved cell lymphoma; stage IV adult diffuse mixed cell lymphoma; stage IV adult diffuse large cell lymphoma; stage IV adult immunoblastic large cell lymphoma; stage IV adult lymphoblastic lymphoma; stage IV adult Burkitt lymphoma; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; recurrent adult diffuse small cleaved cell lymphoma; recurrent adult diffuse mixed cell lymphoma; recurrent adult diffuse large cell lymphoma; recurrent adult immunoblastic large cell lymphoma; recurrent adult lymphoblastic lymphoma; recurrent adult Burkitt lymphoma; stage I mantle cell lymphoma; contiguous stage II grade 1 follicular lymphoma; contiguous stage II grade 2 follicular lymphoma; contiguous stage II grade 3 follicular lymphoma; contiguous stage II adult diffuse small cleaved cell lymphoma; contiguous stage II mantle cell lymphoma; contiguous stage II adult diffuse mixed cell lymphoma; contiguous stage II adult immunoblastic large cell lymphoma; contiguous stage II adult diffuse large cell lymphoma; contiguous stage II adult Burkitt lymphoma; contiguous stage II adult lymphoblastic lymphoma; noncontiguous stage II grade 1 follicular lymphoma; noncontiguous stage II grade 2 follicular lymphoma; noncontiguous stage II grade 3 follicular lymphoma; noncontiguous stage II adult diffuse small cleaved cell lymphoma; noncontiguous stage II mantle cell lymphoma; noncontiguous stage II adult diffuse mixed cell lymphoma; noncontiguous stage II adult immunoblastic large cell lymphoma; noncontiguous stage II adult diffuse large cell lymphoma; noncontiguous stage II adult Burkitt lymphoma; noncontiguous stage II adult lymphoblastic lymphoma; stage III mantle cell lymphoma; stage IV mantle cell lymphoma; recurrent mantle cell lymphoma; noncontiguous stage II small lymphocytic lymphoma; noncontiguous stage II marginal zone lymphoma; recurrent marginal zone lymphoma; recurrent small lymphocytic lymphoma; stage I marginal zone lymphoma; stage I small lymphocytic lymphoma; stage III small lymphocytic lymphoma; stage III marginal zone lymphoma; stage IV small lymphocytic lymphoma; stage IV marginal zone lymphoma; contiguous stage II marginal zone lymphoma; contiguous stage II small lymphocytic lymphoma; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; nodal marginal zone B-cell lymphoma; splenic marginal zone lymphoma
MeSH Terms: conditions — Lymphoma; Lymphoma, Follicular; Lymphoma, Non-Hodgkin; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Large-Cell, Immunoblastic; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Burkitt Lymphoma; Lymphoma, Mantle-Cell; Lymphoma, B-Cell, Marginal Zone; Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Interleukin-12 Subunit p35; Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Biological: recombinant interleukin-12
Biological: rituximab

SUMMARY:
RATIONALE: Interleukin-12 may stimulate a person's white blood cells to kill lymphoma cells. Monoclonal antibodies, such as rituximab, can locate cancer cells and either kill them or deliver cancer-killing substances to them without harming normal cells.

PURPOSE: Phase I trial to study the effectiveness of interleukin-12 plus rituximab in treating patients who have non-Hodgkin's lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the optimal immunological dose of interleukin-12 and rituximab when administered in combination in patients with non-Hodgkin's lymphoma. II. Determine the toxicities associated with this regimen in this patient population. III. Assess the pharmacodynamics of this regimen in these patients. IV. Document observed clinical response to this regimen in these patients.

OUTLINE: This is a dose escalation study of interleukin-12. Patients receive rituximab IV on days 1, 8, 15, and 22. The first cohort of patients receives interleukin-12 SC twice weekly beginning on day 29. Subsequent cohorts receive interleukin-12 SC twice weekly beginning on day 16. Patients with stable or responding disease may continue treatment with interleukin-12 twice weekly for up to 24 weeks or until disease progression. Cohorts of 6-9 patients receive escalating doses of interleukin-12 until the optimal immunological dose is determined. The optimal immunological dose is defined as the dose preceding that at which 2 of 6 or 2 of 9 patients experience dose limiting toxicities or the dose at which there is a maximal increase in gamma interferon, inducible protein-10 (IP-10) and immune cell infiltration into the lymphoma (whichever dose is lower). Following initial dose escalation, 2 additional cohorts of 6 patients receive a fixed dose of interleukin-12 SC twice weekly beginning on day 2. Patients are followed every 3 months for the first year, and then every 6 months for the next 4 years or until disease progression.

PROJECTED ACCRUAL: A maximum of 45 patients will be accrued for this study within 12-13 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed CD20+ B-cell non-Hodgkin's lymphoma No relapsed intermediate or high grade disease eligible for bone marrow or stem cell transplant Intermediate or high grade disease must have received a prior anthracycline containing regimen Low grade disease (with or without prior therapy) felt to be incurable with standard therapy allowed No CNS involvement by lymphoma A new classification scheme for adult non-Hodgkin's lymphoma has been adopted by PDQ. The terminology of "indolent" or "aggressive" lymphoma will replace the former terminology of "low", "intermediate", or "high" grade lymphoma. However, this protocol uses the former terminology.

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: ECOG 0-1 Life expectancy: At least 12 weeks Hematopoietic: Absolute neutrophil count at least 1,500/mm3 Platelet count at least 75,000/mm3 Hemoglobin at least 10 g/dL Hepatic: Bilirubin no greater than 3 times upper limit of normal (ULN) AST/ALT less than 3 times ULN Renal: Creatinine no greater than 2 times ULN Cardiovascular: No New York Heart Association class III or IV heart disease No history of angina Other: Not pregnant or nursing Negative pregnancy test Fertile patients must use effective contraception HIV negative No uncontrolled infection No autoimmune related phenomena No peptic ulcer disease

PRIOR CONCURRENT THERAPY: Biologic therapy: At least 12 months since prior rituximab No prior interleukin-12 No other concurrent immunotherapy Chemotherapy: See Disease Characteristics No prior fludarabine or 2-chlorodeoxyadenosine unless CD4 count normal Recovered from prior chemotherapy No concurrent chemotherapy Endocrine therapy: No concurrent steroid therapy Radiotherapy: No concurrent radiotherapy Surgery: Not specified

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1999-10; Primary Completion 2003-06 (Actual); Study Completion 2003-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen M. Ansell, MD, PhD, Study Chair — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

REFERENCES:
- [Result] Ansell SM, Witzig TE, Kurtin PJ, Sloan JA, Jelinek DF, Howell KG, Markovic SN, Habermann TM, Klee GG, Atherton PJ, Erlichman C. Phase 1 study of interleukin-12 in combination with rituximab in patients with B-cell non-Hodgkin lymphoma. Blood. 2002 Jan 1;99(1):67-74. doi: 10.1182/blood.v99.1.67. PMID 11756154